CLINICAL TRIAL: NCT04371237
Title: Accelerating Post-exercise Muscle Glycogen Resynthesis in Humans: Impact of Combined Nutrient Intake and Intermittent Pneumatic Compression or Heat Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1723
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Muscle Recovery; Muscle Soreness; Glycogen Depletion
Keywords: muscle glycogen; glycogen replenishment; muscle recovery; intermittent pneumatic compression; IPC; heat therapy
MeSH Terms: conditions — Myalgia; Hyperthermia | interventions — Diathermy; Eating; Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent pneumatic compression (Experimental): IPC sleeve device on leg
  Interventions: Device: Compression sleeve; Other: Glycogen-depleting exercise session; Other: Nutrient Intake (beverage); Procedure: Skeletal muscle biopsy
- Heat therapy (Experimental): Custom water-circulating garment on leg
  Interventions: Device: Heat therapy; Other: Glycogen-depleting exercise session; Other: Nutrient Intake (beverage); Procedure: Skeletal muscle biopsy

INTERVENTIONS:
Device: Compression sleeve — From foot to hip/groin on both legs with only 1 leg connected to pneumatic pump for 1 hour
  Other Names: IPC
  Arms: Intermittent pneumatic compression
Device: Heat therapy — Custom leg garment with one leg heated by circulating hot water approx 40 degrees C, the other leg approx 32 degrees C (thermoneutral) for 1 hour
  Arms: Heat therapy
Other: Glycogen-depleting exercise session — Prolonged intermittent high intensity running (LIST protocol)
Other: Nutrient Intake (beverage) — Post-exercise, all participants will receive a beverage containing 1.0 g/kg carbohydrate and 0.3 g/kg protein from the mixture of Gatorade Recover Protein Shake and Gatorade Thirst Quencher
Procedure: Skeletal muscle biopsy — Vastus lateralis muscle in the lower thigh will be obtained by the percutaneous needle technique

SUMMARY:
To determine if modalities designed to improve blood flow combined with post-exercise nutrient intake will improve replenishment of muscle glycogen better than nutrient intake alone. A secondary objective is to compare the effectiveness of heat therapy and intermittent pneumatic compression on glycogen replenishment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be male and female participants in good health
2. 18-35 years of age
3. Currently performing cardiovascular or intermittent exercise at a moderate to high intensity at least 5 days per week for 60 minutes or longer per day.
4. Understanding of the procedures to be undertaken as part of the study
5. Willingness to participate in exercise testing and follow instructions provided by the experimenter
6. Informed, voluntary, written consent to participate in the study

Exclusion Criteria:

1. History of deep vein thrombosis
2. Obesity (BMI > 30 kg/m2)
3. Hypertension (resting SBP > 140/90 mmHg)
4. Smoking
5. Pregnant, planning to become pregnant, or lactating
6. Supplements containing antioxidants including vitamin C and E and N-acetyl cysteine
7. Any medication
8. Lactose intolerance
9. Participation in another study within the previous 30 days or in a PepsiCo funded study within the past 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Rate of glycogen resynthesis | Change from baseline to 1.5 hrs and 3.5 hrs post exercise bout. Biopsy 1 post-exercise pre nutrient intake 1 and compression (IPC) or heat, biopsy 2 post compression or heat, pre-nutrition intake 2, biopsy 3 at 210 min. Higher rate is better.
  Leg skeletal muscle glycogen level assessment using assay kit
Muscle functional recovery: Skeletal muscle function | Change from pre-exercise to post-exercise and prior to biopsies and treatments, and 24 hours post exercise. Less fatigue is better.
  Work fatigue (%) of the knee extensors measured using an isokinetic dynamometer
Muscle functional recovery: Perceived muscle soreness | Change from pre-exercise to post-exercise and prior to biopsies and treatments, and 24 hours post exercise. Less soreness is better.
  Knee extensor muscle soreness on a visual analog scale (VAS) of 100 mm after stepping on and off a 40 cm (female) or 45 cm (male) box three times

SECONDARY OUTCOMES:
mRNA expression of genes involved in regulation of glucose and glycogen metabolism and muscle functional recovery | Change from baseline to 1.5 hours and 3.5 hours post exercise bout. Biopsy 1 post-exercise pre- nutrient intake 1 and compression (IPC) or heat, biopsy 2 post compression or heat and pre- nutrition intake 2, biopsy 3 at 210 min. Higher expression better.
  Leg skeletal muscle fiber analysis determined using RT-PCR (Real-time polymerase chain reaction)
Serum insulin | Change from post exercise at same time as biopsy 1 (Time 0), biopsy 2 (1.5 hrs) and biopsy 3 (3.5 hrs)
  Blood test using ELISA kit
Serum Glucose | Change from post exercise at same time as biopsy 1 (Time 0), biopsy 2 (1.5 hrs) and biopsy 3 (3.5 hrs
  Blood test using ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Roseguini, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, Department of Health & Kinesiology, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No